CLINICAL TRIAL: NCT04399889
Title: Pilot Study of Safety and Efficacy of Cord Tissue Derived Mesenchymal Stromal Cells (hCT-MSC) in COVID-19 Related Acute Respiratory Distress Syndrome (ARDS)
Brief Title: hCT-MSCs for COVID19 ARDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Jerome S. Harris Distinguished Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00105410
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: COVID; Corona Virus Infection; COVID19
Keywords: COVID; Coronavirus infection; COVID19; Covid ARDS; Acute Respiratory Distress Syndrome; ARDS
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open Label infusion of hCT-MSC (Experimental): The first 10 consecutive patients will all receive investigational product.
  Interventions: Biological: Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University.
- Randomized infusion of hCT-MSC (Experimental): An interim analysis, for safety will be conducted and reviewed by the Data Safety and Monitoring Board (DSMB) after the first 10 patients have completed treatment and reached the 28 day endpoint. If there are no safety concerns, the trial will proceed with enrollment on the phase 2 portion of the study where the subsequent 40 patients will be randomized in a 1:1 fashion between treatment with MSCs and placebo. The investigational product will be further randomized to the MSCs manufactured by Duke or University of Miami. These products are considered to be comparable.
  Interventions: Biological: Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University.
- Randomized infusion of Placebo (Placebo Comparator): An interim analysis, for safety will be conducted and reviewed by the Data Safety and Monitoring Board (DSMB) after the first 10 patients have completed treatment and reached the 28 day endpoint. If there are no safety concerns, the trial will proceed with enrollment on the phase 2 portion of the study where the subsequent 40 patients will be randomized in a 1:1 fashion between treatment with MSCs and placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University. — Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University or University of Miami.
  Other Names: hCT-MSC
  Arms: Open Label infusion of hCT-MSC; Randomized infusion of hCT-MSC
Other: Placebo — Placebo will be comprised of 40-80 mL of Plasmalyte-A + 1% Human Serum Albumin (HAS) prepared in an identical container to the one used for cell administration. The placebo product will undergo the same process of sterility testing including release inspection, transport and product custodian.
  Arms: Randomized infusion of Placebo

SUMMARY:
This is a 50 patient, Phase 1/2a multi-center pilot study to test the safety and to describe the preliminary efficacy of intravenous administration of allogenic human cord tissue mesenchymal stromal cells (hCT-MSC) as an investigational agent, under U.S. INDs 19968 (Duke) and 19937 (U Miami) to patients with acute respiratory distress syndrome (ARDS) due to COVID-19 infection (COVID-ARDS). The first 10 consecutive patients will receive investigational MSCs manufactured by Duke. In the second phase of the study, 40 additional patients will be randomized to receive placebo or investigational MSCs manufactured by Duke or University of Miami.

Patients will be eligible for infusion of 3 daily consecutive doses of hCT-MSC or placebo if they have a confirmed diagnosis of COVID-19 and meet clinical and radiographic criteria for ARDS.

Results from the first 10 patients will be compared with concurrent outcomes utilizing standard of care treatments in participating hospitals and in published reports in the medical literature. Results from the additional 40 patients will be combined with the first 10 and analyzed. The trial is relying on focused eligibility of the participants (patients with ARDS), single cohort with short trial time (4 weeks), and simple assessment of clinical outcome (survival, improvement of ARDS). This is a sequential design in the sense that after the first 10 patients are evaluated a decision will be made by the PIs and the Data Safety Monitoring Board whether to proceed with the exploratory randomized portion of the study.

DETAILED DESCRIPTION:
This is a 50 patient, Phase 1/2a multi-center pilot study to test the safety and to describe the preliminary efficacy of intravenous administration of allogenic human cord tissue mesenchymal stromal cells (hCT- MSC) as an investigational agent, under U.S. INDs 19968 (Duke) and 19937 (U Miami) to patients with acute respiratory distress syndrome (ARDS) due to COVID-19 infection (COVID-ARDS). Patients will be eligible for treatment with 3 daily consecutive doses of hCT-MSC at 1 million cells/kg (max dose 100 million cells) in the phase 1 portion of the study or a fixed dose of 100 million cells daily x 3 days, 12-36 hours apart in the phase 2 portion of the study, if they have a confirmed diagnosis of COVID-19 and meet clinical and radiographic criteria for ARDS. The primary endpoint is short-term safety of hCT-MSC infusions given on this schedule. The key secondary endpoints are 28 day survival, an increase in PaO2/FiO2 ratio by 50% at 96 hours, days to hospital discharge to home or rehab, and number of days requiring mechanical or non-invasive ventilation or high flow nasal cannula.

The study will be executed in two phases. The first 10 consecutive patients will all receive investigational product. The second part of the study is a randomized, controlled trial in 40 additional patients. The overall aim of the study is to establish safety and to gain critical information as to whether patients with COVID-ARDS will benefit from MSC infusions. Results from the first 10 patients will be compared with concurrent outcomes utilizing standard of care treatments in participating hospitals and in published reports in the medical literature. Results from the additional 40 patients will be analyzed as a randomized placebo control trial. The trial is relying on focused eligibility of the participants (patients with ARDS), single cohort with short trial time (4 weeks), and simple assessment of clinical outcome (survival, improvement of ARDS). This is a sequential design in the sense that after the first 10 patients are evaluated a decision will be made by the PIs and the Data Safety Monitoring Board whether to proceed with the exploratory randomized portion of the study.

The MSCs are manufactured from allogeneic cord tissue donated to the Carolinas Cord Blood Bank (CCBB) at Duke University. The CCBB is an FDA licensed public cord blood bank (licensed name DUCORD). Cord tissue is donated by mothers delivering healthy term male babies by Cesarean section, after written informed consent from the newborn infant's mother. Full donor screening and testing is performed in accordance with regulatory requirements (21CFR 1271). The hCT-MSCs will be manufactured in the Marcus Center for Cellular Cures in the Robertson GMP Cell Manufacturing Laboratory and the Clinical Research Cell Manufacturing Program (CRCMP) laboratory, Interdisciplinary Stem Cell Institute (ISCI), Miller School of Medicine, University of Miami. These hCT-MSCs are already being utilized in clinical trials to treat pediatric patients with autism spectrum disorder (IND 17313), cerebral palsy (IND 17921), hypoxic ischemic encephalopathy (IND 17313) and adults with osteoarthritis of the knee (IND18414). To date, over 210 doses of cells have been delivered to patients on these clinical trials with an excellent safety profile. At University of Miami, hCT-MSCs are used in the clinical trial to evaluate cytokine suppression in patients with chronic inflammation due to metabolic syndrome (IND 17324), 12 subjects in the pilot phase of the study had completed the dose without any treatment emergence SAE.

The rationale for using this approach for patients infected with COVID-19 is that ARDS, the rate-limiting complication impacting survival, is caused, at least in part, by a cytokine release syndrome (CRS) which results is severe immune dysregulation. Involved cytokines include IL-6, IL-8, IL-10, THP-1M, TNF-alpha, and others. MSCs have strong anti-inflammatory and immune-modulatory activities without apparent toxicity or further immunosuppression. Approximately 3-5 % of patients with COVID-19 develop ARDS which carries a very high mortality rate (30-60%) due to multi-system organ failure. Effective treatment of ARDS, the most feared complication of COVID-19, may convert the COVID-19 pandemic into a more manageable "flu-like" illness that every American is expected to experience, and most will survive, on an annual basis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or legally authorized representative (LAR) must have the ability to understand and the willingness to provide a signed and dated informed consent form.
2. Age 18 years and over
3. The patient agrees to use adequate contraception for the duration of the treatment protocol and for 6 months post treatment.
4. Positive RT- PCR testing for COVID-19 nucleic acid using nasopharyngeal swabbing or any other site
5. Patient meets ARDS criteria and is on non-invasive or mechanical ventilation or high flow nasal cannula

   1. bilateral opacities on chest imaging consistent with pulmonary edema
   2. A need for positive pressure ventilation or high flow nasal cannula
   3. PaO2/FiO2 ratio ≤ 300 mmHg by arterial blood gas or SpO2/FiO2 imputation.
   4. Infiltrates not fully explained by cardiac failure or fluid overload in the physician's best clinical judgement
6. Subjects requiring dialysis as a result of a COVID-19 infection will not be excluded.

Exclusion Criteria:

1. Evidence of multiorgan failure involving one or more organs, excluding the lungs as defined below:

   1. Presence of shock, defined as MAP < 65 mmHg with signs of peripheral hypoperfusion, or continuous infusion of 2 or more vasopressor or inotrope agents to maintain MAP ≥ 65 mmHg.
   2. Serum bilirubin > 10 mg/dl
   3. Platelet count < 50,000/ml
   4. Subjects requiring dialysis as a result of anything other than a COVID-19 infection will be excluded
2. Evidence of acquired or congenital immunodeficiency (due to immunosuppressive therapy excluding steroid use for treatment of COVID-19 acute respiratory failure, HIV, previous treatment for cancer, etc.)
3. History of metastatic cancer diagnosis or treatment in the past 1 year
4. History of previous treatments with MSCs or other cell therapies
5. Patient is co-enrolled in any other IND-sponsored clinical trials for COVID-19 or ARDs. Drugs that are administered under emergency use authorizations (EUA) by the FDA are permitted.
6. Evidence of pregnancy or lactation
7. Moribund patient not expected to survive >24 hours
8. Unable/unwilling to deliver lung protective ventilation
9. Patient is receiving Extracorporeal Membrane Oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke Health; Lingye Chen, MD, Principal Investigator — Duke Health
Locations (5):
- United States (5):
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - New York Medical College, Valhalla, New York
  - Duke Hospital, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Infusion of hCT-MSC: The first 10 consecutive patients all received 3 daily consecutive doses of hCT-MSC at a dose of 1 million cells/kg (maximum 100 million cells).
  Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University.: Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University or University of Miami.
- Randomized Infusion of hCT-MSC: Randomized to 3 daily consecutive doses of hCT-MSC at a dose of 100 million cells.
  Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University.: Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University or University of Miami.
- Randomized Infusion of Placebo: Randomized to 3 daily consecutive infusions of placebo.
  Placebo: Placebo will be comprised of 40-80 mL of Plasmalyte-A + 1% Human Serum Albumin (HAS) prepared in an identical container to the one used for cell administration. The placebo product will undergo the same process of sterility testing including release inspection, transport and product custodian.
Period: Overall Study
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Started | 10 | 1 | 1
Completed | 5 | 0 | 0
Not Completed | 5 | 1 | 1
Not completed — Death | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo | Total
Number analyzed (Participants) | 10 | 1 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (12.3) | 72 (0) | 62 (0) | 63.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 0 | 7
  Male | 3 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 7 | 1 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 0 | 2
  White | 6 | 1 | 1 | 8
  Other | 2 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 1 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Infusion Reactions
Description: Number of infusion reactions measured by any one of the following: fever, anaphylaxis, rash, hypertension, hypotension, tachycardia, nausea, vomiting, or any other new or worsening symptoms associated with the infusion.
Time Frame: 24 hours
Measure: Number; unit: infusion reactions
Groups:
- Open Label Infusion of hCT-MSC: The first 10 consecutive patients all received 3 daily consecutive doses of hCT-MSC at a dose of 1 million cells/kg.
  Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University.: Human cord tissue mesenchymal stromal cells (hCT-MSC) manufactured by Duke University or University of Miami.
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 10 | 1 | 1
infusion reactions | 0 | 0 | 0

2. Primary Outcome: Number of Delayed Reactions
Description: Number of later reactions attributed to the investigational product as measured by any one of the following: rash, infection, allergic reaction, or any other delayed symptoms associated with infusion of the investigational product.
Time Frame: 28 days
Measure: Number; unit: delayed reactions
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 10 | 1 | 1
delayed reactions | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Formation of New Anti-HLA Antibodies
Description: Number of participants who form new anti-HLA antibodies as measured by an antibody screen test at 28 days post first infusion of the investigational product.
Time Frame: 28 days
Population: Data not collected on eight participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 4 | 0 | 0
Participants | 1 | 0 | 0

4. Secondary Outcome: Time to Recovery
Description: Time to recovery, defined as discharge from the hospital (alive) or remaining in the hospital without the need for supplemental oxygen or other COVID-related medical care.
Time Frame: up to 90 days
Population: Participants who recovered.
Measure: Median (Full Range); unit: days
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 5 | 0 | 0
days | 18 [7 to 39] |  |

5. Secondary Outcome: Number of Participants With an Increase in PaO2/FiO2 Ratio
Description: Increase in PaO2/FiO2 ratio by 50% by Day 4 (96 hours after first infusion). PaO2/FiO2 may be calculated from an arterial blood gas or imputed from the SpO2/FiO2 table.
Time Frame: 4 days after MSCs
Population: Data not collected on eight participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 4 | 0 | 0
Participants | 0 |  |

6. Secondary Outcome: Days to Hospital Discharge to Home
Description: The number of days from hospitalization to discharge to home.
Time Frame: 90 days
Population: Participants who were discharged to home.
Measure: Median (Full Range); unit: days
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 3 | 0 | 0
days | 18 [8 to 18] |  |

7. Secondary Outcome: Number of Ventilator Free Days
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 10 | 1 | 1
days | 25.5 [0 to 80] | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Number of Oxygen-free Days
Description: Number of oxygen-free days defined as: 0 if the subject dies within 28 days of supplemental oxygen, 28-x if successfully liberated from supplemental oxygen x days after initiation, and 0 if the subject receives supplemental oxygen for > 28 days.
Time Frame: 28 days
Population: Data not collected on one participant.
Measure: Median (Full Range); unit: days
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 9 | 1 | 1
days | 0 [0 to 21] | 0 [0 to 0] | 0 [0 to 0]

9. Secondary Outcome: Number of Screened Patients Who Are Enrolled and Randomized
Time Frame: 90 days
Population: Open Label infusion of hCT-MSC participants were not randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
Number analyzed (Participants) | 0 | 1 | 1
Participants |  | 1 | 1

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Open Label Infusion of hCT-MSC | Randomized Infusion of hCT-MSC | Randomized Infusion of Placebo
All-Cause Mortality (participants affected / at risk) | 5/10 | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 6/10 | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 4/10 | 0/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Infusion of hCT-MSC (N=10) | Randomized Infusion of hCT-MSC (N=1) | Randomized Infusion of Placebo (N=1)
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1
Death NOS (General disorders) | 2 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Infusion of hCT-MSC (N=10) | Randomized Infusion of hCT-MSC (N=1) | Randomized Infusion of Placebo (N=1)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Fever (General disorders) | 2 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04399889/Prot_SAP_000.pdf